CLINICAL TRIAL: NCT01147523
Title: The Effect of Spironolactone and Vitamin E Versus Vitamin E on Serum Adipocytokines Levels in Patients With Biopsy-proven Nonalcoholic Fatty Liver Disease-A Phase II Study
Brief Title: Effect of Spironolactone and Vitamin E in Patients With Nonalcoholic Fatty Liver Disease
Acronym: NAFLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Stergios A. Polyzos, Dr, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PolyzosKountouras
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Fatty Liver; Steatohepatitis
Keywords: nonalcoholic fatty liver disease; nonalcoholic steatohepatitis; adipokines; spironolactone; vitamin E; adiponectin; visfatin; leptin; resistin; TNF-alpha; IL-6; IL-1
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease | interventions — Spironolactone; Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vitamin E (Experimental): Vitamin E, capsules 400 mg daily, for 52 weeks
  Interventions: Drug: Spironolactone/Vitamin E

INTERVENTIONS:
Drug: Spironolactone/Vitamin E — Spironolactone, tablets, 25 mg daily plus Vitamin E, capsules, 400 mg daily, for 52 weeks
  Other Names: Aldactone tab 25; Eviol caps 100

SUMMARY:
The primary aim of the study is the effect of spironolactone and vitamin E versus vitamin E on serum levels of adipokines 52 weeks post-treatment.

DETAILED DESCRIPTION:
Unlike other chronic liver diseases (e.g., hepatitis C), there are no effective treatment strategy for NAFLD. Currently, the management of NAFLD includes modification of underlying risk factors, detection of patients that have progressed to cirrhosis, management of cirrhosis-related morbidity and transplantation in patients with end-stage liver disease. Diet, exercise, bariatric surgery and pharmacologic treatment, including weight loss agents, insulin sensitizers, lipid-lowering agents, ursodeoxycholic acid and vitamin E have been investigated with some promising results.

The renin-angiotensin-aldosterone system (RAAS) has been implicated in the pathogenesis of insulin resistance (IR) and nonalcoholic fatty liver disease (NAFLD). Recently, low-dose (25-50 mg/day) aldosterone antagonists in patients with heart failure diminish mortality, possibly by reducing cardiac and vascular fibrosis. Moreover, the beneficial effect of spironolactone in a mouse model with diet-induced diabetes and NAFLD has been reported. However, to our knowledge, the role of spironolactone in NAFLD patients has not been investigated yet.

The primary aim of the study is the effect of spironolactone and vitamin E versus vitamin E on serum levels of adipokines 52 weeks post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Bright liver on ultrasound imaging and increased liver function tests for at least 6 months before liver biopsy
* Biopsy-proven NAFLD (either NAFL or NASH) according to NAFLD Activity Score (NAS)

Exclusion Criteria:

* Ethanol consumption more than 20 g/day
* Known intolerance to spironolactone or vitamin E
* History of liver disease (chronic viral hepatitis, autoimmune hepatitis, drug-induced liver disease, primary biliary cirrhosis, hemochromatosis, Wilson's disease and α1-antitrypsin deficiency)
* Previous exposure to hepatotoxic drugs
* Spironolactone or vitamin E administration within one year before screening
* Type I Diabetes Mellitus
* Pancreatitis
* Uncontrolled hypothyroidism or hyperthyroidism
* Adrenal Insufficiency
* Renal Failure
* Cancer
* Pregnancy

Exclusion criteria were generally the same as those proposed for PIVENS trial design with two modifications: a) known intolerance to spironolactone as an exclusion criterion and b) the inclusion of patients with T2DM not receiving thiazolidinediones or insulin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Serum adipocytokines levels | 52 weeks
  Adiponectin; visfatin; leptin; resistin; omentin; vaspin; RBP4; TNF-alpha, IL-6; IL-1

SECONDARY OUTCOMES:
Serum homocysteine levels | 52 weeks
  Homocysteine; vitamin B12; folate
Liver histology | 52 weeks
  Repeat biopsy, if patients provide their consent
Insulin resistance | 52 weeks
  Serum insulin; serum glucose; HOMA and QUICKI indexes
Hormonal profile | 52 weeks
  DHEAS; testosterone; estradiol; TSH; free T4; cortisol (serum levels)
Serum biochemistry | 52 weeks
  ALT; AST; ggt; Potassium; Sodium; urea; creatinin; cholesterol; triglycerides; HDL; LDL
Reactive Oxygen Metabolites (ROMs) | 52 weeks
  Serum dROMs leves

CONTACTS AND LOCATIONS:
Overall Officials: Stergios A Polyzos, MD, MSc, Principal Investigator — Second Medical Clinic, Medical School, Aristotle University of Thessaloniki, Ippokration Hospital, Thessaloniki, Greece; Jannis Kountouras, MD, Prof, Study Chair — Second Medical Clinic, Medical School, Aristotle University of Thessaloniki, Ippokration Hospital, Thessaloniki, Greece; Efthimia Zafeiriadou, MD, PhD, Study Director — Department of Radiology, Ippokration Hospital, Thessaloniki, Greece; Kalliopi Patsiaoura, MD, PhD, Study Director — Department of Pathology, Ippokration Hospital, Thessaloniki, Greece; Evangelia Katsiki, MD, Study Director — Department of Pathology, Ippokration Hospital, Thessaloniki, Greece; Aristidis Slavakis, MD, MSc, Study Director — Department of Biochemistry, Ippokration Hospital, Thessaloniki, Greece
Locations (1):
- Second Medical Clinic, Medical School, Aristotle University of Thessaloniki, Ippokration Hospital, Thessaloniki, Thessaloniki, Greece

REFERENCES:
- [Background] Polyzos SA, Kountouras J, Zavos C. Nonalcoholic fatty liver disease: the pathogenetic roles of insulin resistance and adipocytokines. Curr Mol Med. 2009 Apr;9(3):299-314. doi: 10.2174/156652409787847191. PMID 19355912
- [Background] Polyzos SA, Kountouras J, Zavos C. Insulin resistance and therapy: cross-talk between phosphatidylinositol-3 kinase and mitogen-activated protein kinase pathways. Med Hypotheses. 2009 May;72(5):610. doi: 10.1016/j.mehy.2008.12.019. Epub 2009 Jan 21. No abstract available. PMID 19162411
- [Background] Polyzos SA, Kountouras J, Zavos Ch. The multi-hit process and the antagonistic roles of tumor necrosis factor-alpha and adiponectin in non alcoholic fatty liver disease. Hippokratia. 2009 Apr;13(2):127; author reply 128. No abstract available. PMID 19561788
- [Background] Polyzos SA, Kountouras J, Zavos C. Nonlinear distribution of adiponectin in patients with nonalcoholic fatty liver disease limits its use in linear regression analysis. J Clin Gastroenterol. 2010 Mar;44(3):229-30; author reply 230-1. doi: 10.1097/MCG.0b013e3181b5ce68. No abstract available. PMID 19770674
- [Background] Polyzos SA, Kountouras J, Zavos C, Stergiopoulos C. Adipocytokines in insulin resistance and non-alcoholic fatty liver disease: the two sides of the same coin. Med Hypotheses. 2010 Jun;74(6):1089-90. doi: 10.1016/j.mehy.2009.12.028. Epub 2010 Jan 18. No abstract available. PMID 20080361
- [Background] Polyzos SA, Kountouras J, Zavos C. Adiponectin as a potential therapeutic agent for nonalcoholic steatohepatitis. Hepatol Res. 2010 Apr;40(4):446-7. doi: 10.1111/j.1872-034X.2010.00632.x. No abstract available. PMID 20394676
- [Background] Polyzos SA, Kountouras J, Zavos C, Tsiaousi E. The role of adiponectin in the pathogenesis and treatment of non-alcoholic fatty liver disease. Diabetes Obes Metab. 2010 May;12(5):365-83. doi: 10.1111/j.1463-1326.2009.01176.x. PMID 20415685
- [Background] Polyzos SA, Kountouras J, Zavos C, Deretzi G. The potential adverse role of leptin resistance in nonalcoholic fatty liver disease: a hypothesis based on critical review of the literature. J Clin Gastroenterol. 2011 Jan;45(1):50-4. doi: 10.1097/MCG.0b013e3181ec5c66. PMID 20717042
- [Background] Polyzos SA, Toulis KA, Goulis DG, Zavos C, Kountouras J. Serum total adiponectin in nonalcoholic fatty liver disease: a systematic review and meta-analysis. Metabolism. 2011 Mar;60(3):313-26. doi: 10.1016/j.metabol.2010.09.003. Epub 2010 Oct 30. PMID 21040935
- [Background] Polyzos SA, Kountouras J, Zavos C. Adiponectin in non-alcoholic fatty liver disease treatment: therapeutic perspectives and unresolved dilemmas. Int J Clin Pract. 2011 Mar;65(3):373-4. doi: 10.1111/j.1742-1241.2010.02594.x. No abstract available. PMID 21314876
- [Background] Polyzos SA, Kountouras J, Zavos C, Deretzi G. The association between Helicobacter pylori infection and insulin resistance: a systematic review. Helicobacter. 2011 Apr;16(2):79-88. doi: 10.1111/j.1523-5378.2011.00822.x. PMID 21435084
- [Background] Polyzos SA, Kountouras J, Zavos C, Deretzi G. The potentially dual-faceted nature of fetuin-A in Helicobacter pylori infection and insulin resistance. Clinics (Sao Paulo). 2011;66(5):911-2. doi: 10.1590/s1807-59322011000500031. No abstract available. PMID 21789399
- [Background] Polyzos SA, Kountouras J, Zavos C, Deretzi G. Helicobacter pylori and insulin resistance association: not just a myth, not yet a fact. Saudi J Gastroenterol. 2011 Nov-Dec;17(6):425-6. doi: 10.4103/1319-3767.87190. No abstract available. PMID 22064347
- [Background] Polyzos SA, Kountouras J, Deretzi G, Zavos C, Mantzoros CS. The emerging role of endocrine disruptors in pathogenesis of insulin resistance: a concept implicating nonalcoholic fatty liver disease. Curr Mol Med. 2012 Jan;12(1):68-82. doi: 10.2174/156652412798376161. PMID 22082482
- [Background] Polyzos SA, Kountouras J, Patsiaoura K, Katsiki E, Zafeiriadou E, Deretzi G, Zavos C, Gavalas E, Katsinelos P, Mane V, Slavakis A. Serum homocysteine levels in patients with nonalcoholic fatty liver disease. Ann Hepatol. 2012 Jan-Feb;11(1):68-76. PMID 22166563
- [Background] Polyzos SA, Kountouras J, Patsiaoura K, Katsiki E, Zafeiriadou E, Zavos C, Deretzi G, Tsiaousi E, Slavakis A. Serum vitamin B12 and folate levels in patients with non-alcoholic fatty liver disease. Int J Food Sci Nutr. 2012 Sep;63(6):659-66. doi: 10.3109/09637486.2011.649249. Epub 2012 Jan 9. PMID 22229957
- [Result] Polyzos SA, Kountouras J, Zafeiriadou E, Patsiaoura K, Katsiki E, Deretzi G, Zavos C, Tsarouchas G, Rakitzi P, Slavakis A. Effect of spironolactone and vitamin E on serum metabolic parameters and insulin resistance in patients with nonalcoholic fatty liver disease. J Renin Angiotensin Aldosterone Syst. 2011 Dec;12(4):498-503. doi: 10.1177/1470320311402110. Epub 2011 Mar 24. PMID 21436212
- [Result] Polyzos SA, Kountouras J, Zavos C, Deretzi G. Spironolactone revisited. J Clin Hypertens (Greenwich). 2011 Oct;13(10):783-4. doi: 10.1111/j.1751-7176.2011.00484.x. Epub 2011 Jul 18. No abstract available. PMID 21974769
- [Derived] Polyzos SA, Kountouras J, Anastasilakis AD, Makras P, Hawa G, Sonnleitner L, Missbichler A, Doulberis M, Katsinelos P, Terpos E. Noggin levels in nonalcoholic fatty liver disease: the effect of vitamin E treatment. Hormones (Athens). 2018 Dec;17(4):573-579. doi: 10.1007/s42000-018-0083-8. Epub 2018 Nov 22. PMID 30467685
- [Derived] Polyzos SA, Kountouras J, Mantzoros CS, Polymerou V, Katsinelos P. Effects of combined low-dose spironolactone plus vitamin E vs vitamin E monotherapy on insulin resistance, non-invasive indices of steatosis and fibrosis, and adipokine levels in non-alcoholic fatty liver disease: a randomized controlled trial. Diabetes Obes Metab. 2017 Dec;19(12):1805-1809. doi: 10.1111/dom.12989. Epub 2017 Jul 10. PMID 28452101